CLINICAL TRIAL: NCT07334314
Title: Olfactive Detection of Urothelial Carcinoma by Sniffer Dogs
Acronym: OUAF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9630
Record Dates: First submitted 2025-12-10; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive bladder tumor: Bladder tumor present during cystoscopy and confirmed by pathological examination.
  Interventions: Diagnostic Test: olfactory detection by dogs
- Negative bladder tumor: No bladder tumor on cystoscopy/suspicious lesion but with negative pathological analysis
  Interventions: Diagnostic Test: olfactory detection by dogs

INTERVENTIONS:
Diagnostic Test: olfactory detection by dogs — olfactory detection of urothelial carcinoma of the bladder in a urine sample by dogs

SUMMARY:
The aim of this study is to estimate the sensitivity of olfactory detection of urothelial carcinomas of the bladder in urine samples by assistance dogs trained in this practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years old)
* Subject scheduled for any endourological surgery involving an initial cystoscopy, the most common of which are: transurethral resection of the bladder, transurethral resection of the prostate, internal optical urethrotomy, bladder lithoclast, ureteral stent replacement, ureteroscopy, etc. (non-exhaustive list)
* Subjects for whom a urine sample (for bacteriological or cytological testing) is planned as part of routine practice in the month prior to the procedure
* Subjects affiliated with a health insurance plan or beneficiaries of such a plan

Exclusion Criteria:

* Absence of signed informed consent / inability to provide the subject with informed information (emergency situations, difficulties in understanding the subject, etc.)
* Patient under guardianship, conservatorship, or judicial protection
* History of cancer other than urothelial bladder carcinoma, unless in complete remission for > 5 years
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject scheduled for any endourological surgery involving an initial cystoscopy, the most common of which are: transurethral resection of the bladder, transurethral resection of the prostate, internal optical urethrotomy, bladder lithoclast, ureteral stent replacement, ureteroscopy, etc. (non-exhaustive list).
  Recruitment will take place in the urology department, during the preoperative consultation or during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Assess the sensitivity of olfactory detection of urothelial carcinomas of the bladder in urine samples by assistance dogs trained for this purpose | Day -60 to Day 0

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpitaux Civils de Colmar, Colmar
  - Hôpitaux Universitaires de Strasbourg, Strasbourg